CLINICAL TRIAL: NCT03618810
Title: The Effect, Safety and Pharmacoeconomics of First or Second Level-prophylactic Use of PEG-rhG-CSF in Breast Cancer Patients With Medium-high Risk of Febrile Neutropenia During Chemotherapy
Brief Title: Prophylactic Use of PEG-rhG-CSF in Medium-high Risk of FN in Chemotherapy of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RWS-PEGCSF
Record Dates: First submitted 2018-07-16; First posted 2018-08-07 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Febrile Neutropenia
Keywords: breast cancer; chemotherapy; PEG-rhG-CSF; prophylactic; febrile neutropenia
MeSH Terms: conditions — Febrile Neutropenia; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEGCSF first level prophylactic use: The first level prophylactic use of PEG-rhG-CSF. The Prophylactic use of PEG-rhG-CSF in all cycles of chemotherapy.
  Interventions: Drug: PEGCSF first level prophylactic use
- PEGCSF second level prophylactic use: The second level prophylactic use of PEG-rhG-CSF. The Prophylactic use of PEG-rhG-CSF in the next cycle until FN or 4 grade neutropenia happened.
  Interventions: Drug: PEGCSF second level prophylactic use

INTERVENTIONS:
Drug: PEGCSF first level prophylactic use — 6mg (≥45kg) or 3mg (<45kg) i.h. once 24h after chemotherapy in all cycles of chemotherapy
  Other Names: Xin Rui Bai
  Groups: PEGCSF first level prophylactic use
Drug: PEGCSF second level prophylactic use — 6mg (≥45kg) or 3mg (<45kg) i.h. once 24h after chemotherapy in next cycle if FN or 4 grade neutropenia happened
  Other Names: Xin Rui Bai
  Groups: PEGCSF second level prophylactic use

SUMMARY:
This clinical study is a multiple center, registering and real-world conditional research. The breast cancer patients planning for chemotherapy evaluated with medium-high risk of febrile neutropenia (FN) are recruited, receiving the first level prophylactic use of PEG-rhG-CSF or the second level prophylactic use of PEG-rhG-CSF in at least two cycles of chemotherapy according to real-world clinical judgement and choice by physicians in local cancer center. Comparing real conditional-FN rate, FN-caused hospitalization rate and antibiotic use rate, direct/indirect medical cost.

DETAILED DESCRIPTION:
The breast cancer patients planning for neo-adjuvant/adjuvant chemotherapy evaluated with medium-high risk of febrile neutropenia (FN) according to NCCN and ASCO guideline are recruited, receiving the first level prophylactic use of PEG-rhG-CSF or the second level prophylactic use of PEG-rhG-CSF according to real-world clinical judgement and choice by physicians in local cancer center for at least two cycles of chemotherapy. The primary outcome is FN rate, the second outcomes are rate of 3-4 grade decrease of ANC, FN-caused hospitalization, FN-caused antibiotic use rate, rate of reduction of chemotherapy dose, delay of chemotherapy, safety and pharmacoeconomics.

ELIGIBILITY:
Inclusion Criteria:

1. provision of informed consent
2. stage I-III, invasive breast cancer
3. accept at least 4 cycles of chemotherapy
4. ECOG score 0-2
5. with medium-high risk of FN according to researchers

Exclusion Criteria:

1. accepted stem cell or bone marrow transplant
2. undergoing any other clinical trial
3. uncontrolled infection, temperature≥38℃
4. per-week scheme chemotherapy
5. concurrent with radiotherapy
6. allergic conditions
7. sever organ dysfunction
8. uncontrolled diabetes

Ages: 13 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergoing chemotherapy given by prophylactic PEG-rhG-CSF using for preventing FN.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-20 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
FN rate | assessment at 1 month after the last cycle chemotherapy complete
  rate of febrile neutropenia during all cycles of chemotherapy

SECONDARY OUTCOMES:
rate of 3-4 grade neutropenia | During all cycles of chemotherapy, through study completion, an average of half year
  rate of 3-4 grade decrease of ANC
FN-caused hospitalization | During all cycles of chemotherapy, through study completion, an average of half year
  rate of FN-caused hospitalization
FN-caused antibiotic use rate | During all cycles of chemotherapy, through study completion, an average of half year
  rate of FN-caused antibiotic use
rate of dose reduction | During all cycles of chemotherapy, through study completion, an average of half year
  rate of reduction of chemotherapy dose

CONTACTS AND LOCATIONS:
Overall Officials: Hongjian Yang, MD, Principal Investigator — Zhejiang Cancer Hospital